CLINICAL TRIAL: NCT02126761
Title: A Phase 1, Randomized, Observer Blind, Antigen and Adjuvant Dosage-Finding Study to Evaluate the Safety and Immunogenicity of an Adjuvanted, Trivalent Subunit Influenza Vaccine in Elderly Subjects ≥65 Years of Age
Brief Title: Safety and Immunogenicity of Different Formulations of an Adjuvanted, Trivalent Subunit Influenza Vaccine in Elderly Subjects 65 Years of Age and Above
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seqirus (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V133_01EXP; 2013-005344-29 (EudraCT Number)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2015-12

CONDITIONS: Influenza
Keywords: Influenza; elderly; adjuvant
MeSH Terms: conditions — Influenza, Human | interventions — Antigens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Group 1 (Active Comparator): aTIV
  Interventions: Biological: Adjuvanted, trivalent subunit influenza vaccine
- Group 2 (Experimental): aTIV + 1X MF59
  Interventions: Biological: Adjuvant level modified adjuvanted, trivalent subunit influenza vaccine
- Group 3 (Experimental): aTIV + TIV
  Interventions: Biological: Antigen level modified adjuvanted, trivalent subunit influenza vaccine
- Group 4 (Experimental): aTIV + aTIV
  Interventions: Biological: Antigen and adjuvant level modified adjuvanted, trivalent subunit influenza vaccine
- Group 5 (Active Comparator): aTIV (Left deltoid) Saline (Right deltoid)
  Interventions: Biological: Adjuvanted, trivalent subunit influenza vaccine
- Group 6 (Experimental): aTIV+2X MF59 (Left deltoid) Saline (Right deltoid)
  Interventions: Biological: Adjuvant level modified adjuvanted, trivalent subunit influenza vaccine
- Group 7 (Experimental): aTIV (Left deltoid) aTIV (Right deltoid)
  Interventions: Biological: Antigen and adjuvant level modified adjuvanted, trivalent subunit influenza vaccine

INTERVENTIONS:
Biological: Adjuvanted, trivalent subunit influenza vaccine — Group 1 and group 5 are active comparators; group 5 includes placebo comparator as a second injection in contralateral deltoid
  Arms: Group 1; Group 5
Biological: Adjuvant level modified adjuvanted, trivalent subunit influenza vaccine — Group 2 and group 6 are experimental; group 2 has double dosage of MF59 in a single injection; group 6 has triple dosage of MF59 and includes placebo comparator in contralateral deltoid
  Arms: Group 2; Group 6
Biological: Antigen level modified adjuvanted, trivalent subunit influenza vaccine — Group 3 is experimental with double the usual antigen dosage
  Arms: Group 3
Biological: Antigen and adjuvant level modified adjuvanted, trivalent subunit influenza vaccine — Group 4 and 7 are experimental; group 4 has one injection with double the antigen and adjuvant; group 7 has two injections with double the antigen and adjuvant
  Arms: Group 4; Group 7

SUMMARY:
In this study, the safety and immunogenicity of the current formulation of aTIV will be compared to aTIV-modified formulations in which the dosage of the MF59 adjuvant will be doubled or tripled and/or the dosage of the 3 influenza virus strains will be doubled, in independently-living elderly subjects ≥ 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥65 years of age on the day of screening who are healthy or have chronic illnesses that are stable and well controlled.
2. Subjects assessed as mentally competent, who have given informed consent after the nature of the study has been explained according to local requirements
3. In good health as determined by:

   1. Ability to live independently
   2. Medical history
   3. Physical examination
   4. Clinical judgment of the Investigator
4. Able to understand and comply with all study procedures and visits, and are able to complete an eDiary
5. Individuals who have access to a working telephone and are able to receive periodic telephone calls

Exclusion Criteria:

1. Individuals who have received any type of influenza vaccine (licensed or experimental) within the past 6 months
2. Individuals who have received any other licensed vaccines within 30 days (for inactivated vaccines) or 42 days (for live vaccines) prior to enrollment in this study
3. Individuals who have cancer except for:

   1. Benign localized skin cancer
   2. Localized prostate cancer that has been clinically stable for ≥ 2 years without treatment
   3. Cancer in remission for ≥ 10 years (from end of cancer treatment)
4. Individuals with autoimmune disease (including rheumatoid arthritis)
5. Individuals with diabetes mellitus, type I
6. Individuals with a body mass index (BMI) ≤18 or ≥35.
7. Asthma that is greater than mild in severity and / or has exacerbations more than 2 days per week
8. Congestive heart failure with symptoms as severe as or more severe than dyspnea with short walks or climbing a single flight of stairs (for example, greater than New York Heart Association class 2)
9. History of progressive or severe neurologic disorders including but not limited to multiple sclerosis, Parkinson's disease, Guillain-Barré syndrome, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, epilepsy disorders requiring medication for control, encephalitis, Alzheimer's and CVA
10. Individuals who are hypersensitive to ovalbumin, chicken protein, chicken feathers, influenza viral protein, kanamycin and neomycin sulfate or any other component of the vaccines in study
11. Individuals who have a history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine
12. Individuals who have a known or suspected (or have a high risk of developing) impairment/alteration of immune function resulting from, for example,

    a. Receipt of immunosuppressive therapy (defined as follows) within the past 60 days and/or anticipated to receive immunosuppressive therapy at any point within 21 days of Visit 1.

    i. Cancer chemotherapy/radiotherapy ii. Systemic corticosteroids ( i.e., 15 mg or greater per day of prednisone or equivalent) iii. Chronic use of inhaled/intranasal high potency corticosteroids (budesonide 800 μg per day or fluticasone 750 μg per day) b. Receipt of immunostimulants c. Receipt of parenteral immunoglobulin preparation, blood products and/or plasma derivate within the past 3 months and for the full length of the study d. Suspected or known HIV infection or HIV-related disease
13. Individuals who have a known or suspected history of drug or alcohol abuse
14. Individuals who, within the past 12 months, have had laboratory confirmed influenza disease
15. Individuals who, within the past 30 days have received any investigational agent.
16. Individuals who plan to receive another vaccine within 30 days of receipt of the study vaccination.
17. Individuals who, within the past 14 days, have experienced:

    1. Any acute disease including any worsening of underlying respiratory diseases such as asthma or COPD
    2. Infections requiring systemic antibiotic or antiviral therapy (chronic antibiotic therapy for urinary tract prophylaxis is acceptable)
18. Individuals who are taking part in another clinical study
19. Individuals who are research staff directly involved with the clinical study or family members or household members of research staff. Research staff includes an individual with direct or indirect contact with study subjects, or study site personnel who have access to any study documents containing subject information. This would include receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians, etc.
20. Individuals with behavioral or cognitive impairment or a psychiatric condition that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
21. Vulnerable subjects, e.g. subjects kept in detention, soldiers, employees of the sponsor or a clinical research organization involved in this study
22. Individuals who have any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 196 (Actual)
Dates: Start 2014-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Reactogenicity up to 7 days after vaccination | Days 1-7 post-vaccination
  Safety of aTIV or aTIV-modified formulations
Unsolicited AEs within 28 days after vaccination | Days 1-28 post-vaccination
SAEs, non-scheduled physician visits, unsolicited medically attended AEs, unsolicited AEs leading to study withdrawal, NOCDs, and AESIs from study start to study completion. | Days 1-366 post-vaccination
Seroconversion/significant increase in antibody HI titers; ≥4-fold rise in MN titer 21 days post-vaccination. | Day 22 post-vaccination
  Antibody responses to all three influenza virus vaccine strains, 21days after a dose or doses of aTIV or aTIV-modified formulations, as measured by hemagglutination inhibition (HI) assay and microneutralization (MN) assay.
HI and MN GMT and GMR at baseline and 21 days post-vaccination. | Day 1; Day 22 post-vaccination

SECONDARY OUTCOMES:
Seroconversion/significant increase in antibody HI titers; ≥4-fold rise in MN titer, 7 days and 6 months post-vaccination. | Day 8 and 181 post-vaccination
HI and MN (GMT) 7 days and 6 months post-vaccination. | Day 8 and 181 post-vaccination
  To compare HI and MN responses to a aTIV or aTIV-modified formulations, at 7 days and 6 months post-vaccination.
HI and MN (GMR) 7 days, 21 days, and 6 months post-vaccination. | Day 1, 8, 22, and 181 post-vaccination
Percentage of subjects with HI titers ≥1:40, ≥1:110, ≥1:160, and ≥1:330 7 days, 21 days, and 6 months post-vaccination. | Day 8, 22, and 181 post-vaccination
  To compare antibody responses in subjects receiving aTIV-modified formulations in a single intramuscular injection (in one deltoid) to two intramuscular injections (one in each deltoid) at 7 days, 21 days, and 6 months post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- PAREXEL Early Phase Clinical Unit, Berlin, Germany